CLINICAL TRIAL: NCT00865449
Title: Role of Renin Angiotensin Blockade in Peritoneal Fibrosis in Peritoneal Dialysis Patients
Brief Title: Spironolactone and Prevention of Peritoneal Fibrosis in Peritoneal Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Magdalena Madero, MD, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08-590
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2009-03

CONDITIONS: End Stage Renal Disease
Keywords: spironolactone; peritoneal fibrosis; peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Peritoneal Fibrosis | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Peritoneal Dialysis patients on aldactone for 6 months
  Interventions: Drug: spironolactone
- 2 (Placebo Comparator): Peritoneal dialysis Patients on the placebo arm for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: spironolactone — 25 mg daily of spironolactone given for 6 months in the peritoneal dialysis patients
  Arms: 1
Drug: Placebo — Placebo, given daily for 6 months to Peritoneal Dialysis Patients
  Arms: 2

SUMMARY:
This is a double blind randomized controlled study to evaluate the effect of aldactone on peritoneal fibrosis on incident peritoneal dialysis patients. The study would include a total of 40 incident peritoneal dialysis patients. Peritoneal biopsy would be made at randomization and 6 months after the intervention to evaluate the effect of renin angiotensin blockade on peritoneal fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Hospitalized for peritoneal catheter placement for peritoneal dialysis

Exclusion Criteria:

* Pregnancy
* Hiperkalemia (K> 5.5meq/l)
* Intolerance to spironolactone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Peritoneal fibrosis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Madero, M.D, Principal Investigator — Instituto Nacional de Cardiologia Ignacio Chavez
Locations (1):
- Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138